CLINICAL TRIAL: NCT00583336
Title: Physician Preference Study of the Utility of ShuntCheck to Detect Cerebrospinal Fluid (CSF) in Patients With Ventriculo-Peritoneal CSF Shunts
Brief Title: Physician Preference Study of ShuntCheck - Madsen
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: NeuroDx Development (Industry)
Collaborators: Boston Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NDX 07-07-0277; 07-07-0277
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: CSF Flow Through the Shunt of a Hydrocephalus Patient

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diagnostic (Experimental)
  Interventions: Device: ShuntCheck

INTERVENTIONS:
Device: ShuntCheck — Thermal dilution test for CSF flow

SUMMARY:
ShuntCheck can be used to detect CSF flow in asymptomatic hydrocephalus patients and can be used to detect no-flow in symptomatic patients with shunt obstruction.

Secondarily, the ShuntCheck test will yield the clearest results when patients are tested sitting up (or alternatively while supine)

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be 0 - 85 years of age, of any race or sex with parent consent for minors
2. Subjects must have a chronically indwelling ventriculo-peritoneal shunt that is palpable along the clavicle.
3. Subjects must be physically stable as determined by the physician.

Exclusion Criteria:

1. Subjects with the presence of an open wound at the shunt site that could interfere with the collection of ShuntCheck data.
2. Subjects unable to lie supine with head elevated 30 degrees or less
3. Subjects who have had shunt surgery within two weeks.
4. Inability or unwillingness of subject to endure the test.
5. Other judgments of the investigator.

Max Age: 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2007-09; Primary Completion 2015-07 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
ShuntCheck result of "Flow Confirmed" for asymptomatic shunted patients tested | Tested in single visit

SECONDARY OUTCOMES:
ShuntCheck result of "Flow Not Confirmed" for symptomatic shunted patients with shunt obstruction | Single visit

CONTACTS AND LOCATIONS:
Overall Officials: Joseph R Madsen, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States